CLINICAL TRIAL: NCT03729960
Title: Cry Management and Awareness Tool (Cool): A Proof of Concept Study to Investigate the Use and Relevance of a Digital Platform for Infant Crying and Fussing
Brief Title: A Proof of Concept Study to Investigate the Use and Relevance of a Digital Platform for Infant Crying and Fussing
Acronym: COOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: Tech Observer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EBB17GC16811_2
Record Dates: First submitted 2018-08-22; First posted 2018-11-05 (Actual); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LENA (Other): Lena device with Fitbit and Cocooncam being optional
  Interventions: Other: LENA recorder

INTERVENTIONS:
Other: LENA recorder — The LENA recorder model# 0121 is a lightweight, pocket-size, rechargeable electronic recorder together with a mobile application to view the data and answer questionnaires
  Other Names: Fitbit, Cool Mobile app,Cocoon Cam

SUMMARY:
Primary: The rating by the primary caregivers on the use and relevance of data provided by the Language ENvironment Analysis (LENA) recorder and their level of engagement due to the content on the Cool mobile app.

Secondary: The rating by the Healthcare Professionals (HCPs) on the use and relevance of data provided by the LENA recorder in their general practice

Exploratory

* Total crying and fussing time captured by the LENA recorder
* Crying and fussing time perceived by the parents
* Vital parameters like heart rate, sleep recorded by the Fitbit used by the primary caregiver during crying and fussing events registered by LENA
* Comments and feedback provided by the primary caregiver on the LENA recorder and the Cool mobile app
* Comments and feedback provided by the HCP on the LENA recorder and the data provided.
* Sleep time recorded by the Cocoon Cam
* Crying time recorded by the Cocoon Cam
* Crying start and end time recorded by the primary caregiver in the COOL app
* Sleep start and end time recorded by the primary caregiver in the COOL app
* Comments and feedback provided by the primary caregiver and HCP on the Cocoon Cam and the activity log for infant cry and sleep including push notifications in the Cocoon Cam app
* Usage data from the Cocoon Cam app

DETAILED DESCRIPTION:
At screening visit, after parent(s)/guardian(s) of potential subjects and/or legal representatives have been informed about the study, they will be requested to sign the informed consent form (ICF) prior to start of the study. After successful signing of the informed consent, the investigator will assess the eligibility of the subjects. If the subject meets all the inclusion and none of the exclusion criteria, the primary caregiver will complete a detailed questionnaire on subject's demographics, birth, family, feeding characteristics and primary caregiver's characteristics. The primary caregiver will be provided the LENA recorder kit and in case consented for Fitbit, they will be provided with the Fitbit. The primary caregiver will need to complete a training period in order to verify subject's primary caregiver's ability to properly connect, operate and upload data using the LENA recorders and uploader. As part of the training period, the primary caregiver will do 1-2 hours of recording using the LENA recorder and successfully upload the data into the LENA cloud server through the internet. Once the study coordinator verifies that the upload is successful, the training and feasibility assessment will be considered as complete and the subject will be considered as enrolled. The primary caregiver of the enrolled subject will be provided access to the COOL mobile app and the recording period will start.

During the recording period, the subject will be using the LENA recorder and will complete a daily questionnaire at the end of each day. At the end of 7 days, the site will perform a phone call and the LENA cry and fuss clock generated from the LENA recorder data for the recorded period will be shared with the primary caregiver through the COOL mobile app. After viewing the cry and fuss clock, the primary caregiver will need to complete a questionnaire on the use of LENA recorder and the content of the COOL mobile app. The primary caregiver will continue using the LENA recorder for the next 7 days. At the end of 14 days, the LENA cry and fuss data for the recorded period will be shared with the primary caregiver and the primary caregiver will need to complete another questionnaire on the use and relevance of the cry and fuss clock and overall relevance of the COOL mobile app. At the end of the recording period, the primary caregiver will schedule an appointment with the PI. If the primary caregiver consents for the use of Fitbit, they will be provided Fitbit to record their vital parameters like heartrate and sleep pattern through the 14 days after enrolment. At the end of study visit, the primary caregiver will discuss the data provided by the LENA recorder and the COOL mobile app with the PI and PI will use the data to explain to the primary care giver if there is any specific cry pattern that could be assessed based on the objective data from LENA. The Primary caregiver and PI will complete a questionnaire each on the use of the data provided by the LENA recorder during their discussion.

For up to 5 subjects in the study, if the primary caregiver consents for the use of Cocoon Cam they will be provided with the Cocoon Cam kit at screening visit. The primary caregiver will need to complete a training period to verify the ability to properly connect, operate and upload data using the LENA recorders and uploader as well as the Cocoon Cam. As part of the training period, the primary caregiver will have to I) perform 1-2 hours of recording using the LENA recorder II) successfully upload the data into the LENA cloud server through the internet, III) use the Cocoon Cam for 1 day, and IV) be able to start using the Cocoon Cam application. Once the study coordinator verifies that the LENA upload is successful and Cocoon Cam set-up is complete, the training and feasibility assessment will be considered as complete and the subject will be considered as enrolled. The primary caregiver of the enrolled subject will be provided access to the COOL mobile app and the recording period will start. During the recording period, in addition to the daily questionnaire, the primary caregiver need to enter cry and sleep time using the COOL app. At the end of 7th day and 14th day, the primary caregiver need to complete questionnaires on the usability of the Cocoon Cam.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 2 to 12 months.
2. Primary caregiver should have reliable access to the internet and a reliable device such as a computer, tablet or smart phone to access the Cool mobile app and able to view the LENA data and complete questionnaires.
3. Primary caregiver should be adequately skilled comfortable in English to read the content in the Cool mobile app and complete questionnaires.
4. Primary caregiver takes care of the child more than 50% of the time.

Exclusion Criteria:

1. Primary caregiver who is not adequately skilled comfortable in English language to read the content in the Cool mobile app and complete questionnaires.
2. Incapability of the primary caregiver to access Cool mobile app through internet.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SBCC Clinic Pte Ltd, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LENA
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LENA
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.77 (2.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 18
  Others | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 20

OUTCOME MEASURES:

1. Primary Outcome: The Rating by the Primary Caregivers on the Use and Relevance of the Cry and Fuss Clock Generated From the LENA Recorder Data and the Rating by the Primary Caregiver on the Level of Engagement Due to the Content on the COOL Mobile App.
Description: Rating by the primary caregiver about the usability and relevance using a 6-point scale [0=Not at all, 5=Yes, very much]; Scale 1 to 4 is subjective to user definition (not defined specifically)
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Groups:
- LENA: Lena device with both Fitbit and Cocooncam being optional
  LENA recorder: The LENA recorder model# 0121 is a lightweight, pocket-size, rechargeable electronic recorder together with a mobile application to view the data and answer questionnaires
Arm/Group | LENA
Number analyzed (Participants) | 20
Participants
  Use and relevance scale 0 - Not at all | 3
  Use and relevance Scale 1 | 1
  Use and relevance Scale 2 | 3
  Use and relevance Scale 3 | 6
  Use and relevance Scale 4 | 7
  Use and relevance Scale 5 - Yes, very much | 0

2. Secondary Outcome: The Rating by the HCPs on the Use and Relevance of Data Provided by the LENA Recorder in Their General Practice.
Description: Rating by the HCP about the use and relevance of the LENA data in general practice using 6 point scale [0=Not at all, 5=Yes, very much], Scale 1 to 4 is subjective to user definition (not defined specifically)
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | LENA
Number analyzed (Participants) | 20
Participants
  Use and relevance scale 0 - Not at all | 0
  Use and relevance Scale 1 | 0
  Use and relevance Scale 2 | 6
  Use and relevance Scale 3 | 6
  Use and relevance Scale 4 | 8
  Use and relevance Scale 5 - Yes, very much | 0

3. Other Pre Specified Outcome: Exploratory Parameter :Total Crying and Fussing Time Captured by the LENA Recorder
Description: Exploratory Parameter : Total daily crying and fussing time captured by the LENA recorder in minutes
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LENA
Number analyzed (Participants) | 20
minutes | 19.6 (30.7)

4. Other Pre Specified Outcome: Exploratory Parameter :Crying and Fussing Time Perceived by the Parents
Description: Daily duration of cry and/or fuss in the scale of :
  <30 mins 30 mins to 1hr >1hr to 3hrs > 3hrs
Time Frame: 2 weeks
Population: The question was asked everyday within the 2 weeks' time frame. Data used to estimate number of participant days over (15 days x 20 participants) 300 participant days for each category of cry. For example, over a period of 15 days (Day 0 to Day 14) equivalent to 2 weeks time frame, the category "<30 mins" was selected 105 times by 20 participants.
Measure: Number; unit: participant days
Units Other Than Participants: participant days
Arm/Group | LENA
Number analyzed (Participants) | 20
Number analyzed (participant days) | 300
participant days
  < 30 mins | 105
  30 mins to 1hr | 86
  >1hr to 3hrs | 82
  >3hrs | 16
  Missing | 11

5. Other Pre Specified Outcome: Usage Time of the Cocoon Cam App by the Primary Caregiver
Description: Usage time (in minutes) of the Cocoon Cam app by the primary caregiver.
Time Frame: 2 weeks
Population: 20 participants enrolled into study, 5 participants enrolled to use cocoon cam app but only 4 had data as 1 had wifi issue connecting to cocoon cam app.
Measure: Mean (Full Range); unit: minutes
Arm/Group | LENA
Number analyzed (Participants) | 5
minutes | 4.1 [0 to 14.4]

6. Other Pre Specified Outcome: To Explore the Usability of Cocoon Cam and Data Captured by the Cocoon Cam App for the HCP in Their Daily Practice
Description: To explore the usability of Cocoon Cam and data captured by the Cocoon Cam app for the HCP in their daily practice. Scale 0 = Not at all, Scale 5 = Yes very much. Scale 1 to 4 is subjective to user definition (not defined specifically)
Time Frame: 2 weeks
Population: 5 participants enrolled to cocoon cam app use but 1 participant had issue with wifi connection so only 4 had data
Measure: Count of Participants; unit: Participants
Arm/Group | LENA
Number analyzed (Participants) | 5
Participants
  Use and relevance scale 0 - Not at all | 1
  Use and relevance Scale 1 | 0
  Use and relevance Scale 2 | 2
  Use and relevance Scale 3 | 2
  Use and relevance Scale 4 | 0
  Use and relevance Scale 5 - Yes, very much | 0

ADVERSE EVENTS:
Time Frame: 15 days (Day 0 to Day 14)
Arm/Group | LENA
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT03729960/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03729960/SAP_001.pdf